CLINICAL TRIAL: NCT05284422
Title: Effect of Ultrasound-guided Insertion of Peripheral Catheters in the Forearm in Complications Incidence.
Brief Title: Effect of Ultrasound-guided Insertion on Peripheral Catheters Related Complications.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PR(AMI)24/2021
Record Dates: First submitted 2022-02-14; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Catheter Related Complication
Keywords: peripheral; ultrasound-guided

STUDY DESIGN:
Intervention Model Description: Participants are assigned to the traditional or ultrasound-guided insertion group
Who Masked: Participant, Care Provider, Investigator
Masking Description: A random list is generated by a computer randomizer program. Sealed numbered envelopes are prepared with study documents and the technique to be performed. Investigators take envelops in consecutive order as long as participants accept to be included in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional technique (Active Comparator): Peripheral venous catheters inserted to the participants in this arm are inserted with a palpation/visualization guided technique in their hand, arm, foot or head.
  Interventions: Procedure: Traditional Peripheral venous catheter insertion
- Ultrasound-guided technique (Experimental): Peripheral venous catheters inserted to the participants in this arm are inserted with an ultrasound-guided technique in their forearm.
  Interventions: Procedure: Ultrasound-guided insertion of a peripheral venous catheter

INTERVENTIONS:
Procedure: Traditional Peripheral venous catheter insertion — Insertion of a short catheter in a peripheral vein with the help of visualization palpation
  Arms: Traditional technique
Procedure: Ultrasound-guided insertion of a peripheral venous catheter — Insertion of a short catheter in a peripheral vein with the help of an ultrasound device
  Arms: Ultrasound-guided technique

SUMMARY:
The purpose of this study is to compare the appearance of complications after the insertion of peripheral venous catheters with two different techniques (traditional and ultrasound-guided).

DETAILED DESCRIPTION:
All patients, whose parents were informed about the study and give written informed consent, will be randomized in a double-blind manner (participant and investigator) in a 1:1 ratio to visualization/palpation or ultrasound-guided peripheral catheter insertion. All participants undergo a 10 days monitoring of the catheter status.

ELIGIBILITY:
Inclusion Criteria:

* Age between 0 and 18 years
* Patients in need of a peripheral venous catheter

Exclusion Criteria:

* Inability of insertion in both forearms (i.e. burnt, amputation)
* Patients in need of a central venous catheter

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 376 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants presenting peripheral catheter insertion-related complications for each intervention | From catheter insertion until the date of documented complication or catheter withdrawal assessed up to 10 days
  Peripheral insertion-related complications: phebitis, infiltration, catheter loss, obstruction

SECONDARY OUTCOMES:
Demographic traits of participants presenting peripheral catheter-related complications | From catheter insertion until the date of documented complication or catheter withdrawal assessed up to 10 days
  Age average (years) and gender (male/female)
The proportion of canalization aspects in peripheral catheter-related complications | From catheter insertion until the date of documented complication or catheter withdrawal assessed up to 10 days
  Catheter size (Ga), operator experience (years), insertion site (hand/forearm/arm/foot/head), insertion ward (PICU/ER)
Number of participants that present immobilization of the limb in both techniques | From catheter insertion until the date of documented complication or catheter withdrawal assessed up to 10 days
  Immobilization of the limb where the peripheral catheter is inserted (Yes/No)
Use of the catheter inserted in participants presenting peripheral catheter-related complications | From catheter insertion until the date of documented complication or catheter withdrawal assessed up to 10 days
  Type of fluid infusion, antibiotic administration (Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The name and location (ward/room) of participants will be accessible to researchers until the peripheral catheter withdrawal.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: From the insertion to the withdrawal of the peripheral venous catheter.
Access Criteria: Investigator will access individual participant data to monitor and register the catheter condition

REFERENCES:
- [Background] Ben Abdelaziz R, Hafsi H, Hajji H, Boudabous H, Ben Chehida A, Mrabet A, Boussetta K, Barsaoui S, Sammoud A, Hamzaoui M, Azzouz H, Tebib N. Peripheral venous catheter complications in children: predisposing factors in a multicenter prospective cohort study. BMC Pediatr. 2017 Dec 19;17(1):208. doi: 10.1186/s12887-017-0965-y. PMID 29258474
- [Background] Carr PJ, Rippey JCR, Cooke ML, Higgins NS, Trevenen M, Foale A, Rickard CM. From insertion to removal: A multicenter survival analysis of an admitted cohort with peripheral intravenous catheters inserted in the emergency department. Infect Control Hosp Epidemiol. 2018 Oct;39(10):1216-1221. doi: 10.1017/ice.2018.190. Epub 2018 Sep 10. PMID 30196798
- [Background] Benkhadra M, Collignon M, Fournel I, Oeuvrard C, Rollin P, Perrin M, Volot F, Girard C. Ultrasound guidance allows faster peripheral IV cannulation in children under 3 years of age with difficult venous access: a prospective randomized study. Paediatr Anaesth. 2012 May;22(5):449-54. doi: 10.1111/j.1460-9592.2012.03830.x. Epub 2012 Mar 12. PMID 22409596
- [Background] Suliman M, Saleh W, Al-Shiekh H, Taan W, AlBashtawy M. The Incidence of Peripheral Intravenous Catheter Phlebitis and Risk Factors among Pediatric Patients. J Pediatr Nurs. 2020 Jan-Feb;50:89-93. doi: 10.1016/j.pedn.2019.11.006. Epub 2019 Nov 27. PMID 31785409
- [Background] Doniger SJ, Ishimine P, Fox JC, Kanegaye JT. Randomized controlled trial of ultrasound-guided peripheral intravenous catheter placement versus traditional techniques in difficult-access pediatric patients. Pediatr Emerg Care. 2009 Mar;25(3):154-9. doi: 10.1097/PEC.0b013e31819a8946. PMID 19262420
- [Background] Indarwati F, Mathew S, Munday J, Keogh S. Incidence of peripheral intravenous catheter failure and complications in paediatric patients: Systematic review and meta analysis. Int J Nurs Stud. 2020 Feb;102:103488. doi: 10.1016/j.ijnurstu.2019.103488. Epub 2019 Nov 26. PMID 31862530
- [Background] Cicolini G, Manzoli L, Simonetti V, Flacco ME, Comparcini D, Capasso L, Di Baldassarre A, Eltaji Elfarouki G. Phlebitis risk varies by peripheral venous catheter site and increases after 96 hours: a large multi-centre prospective study. J Adv Nurs. 2014 Nov;70(11):2539-49. doi: 10.1111/jan.12403. Epub 2014 Mar 31. PMID 24684163
- [Background] Salleras-Duran L, Fuentes-Pumarola C, Bosch-Borras N, Punset-Font X, Sampol-Granes FX. Ultrasound-Guided Peripheral Venous Catheterization in Emergency Services. J Emerg Nurs. 2016 Jul;42(4):338-43. doi: 10.1016/j.jen.2015.11.005. Epub 2016 Mar 4. No abstract available. PMID 26953509
- [Background] Takeshita J, Nakayama Y, Nakajima Y, Sessler DI, Ogawa S, Sawa T, Mizobe T. Optimal site for ultrasound-guided venous catheterisation in paediatric patients: an observational study to investigate predictors for catheterisation success and a randomised controlled study to determine the most successful site. Crit Care. 2015 Jan 20;19(1):15. doi: 10.1186/s13054-014-0733-4. PMID 25600063